CLINICAL TRIAL: NCT00363454
Title: Phase I Pharmacokinetic and Pharmacodynamic, Open-Label, Dose Escalation Study of Triciribine Phosphate Monohydrate (TCN-PM, VD-0002) in Adult Subjects With Metastatic Cancer Which Have Activated Akt Demonstrated by Immunohistochemistry
Brief Title: Phase I Study of Triciribine Phosphate Monohydrate (TCN-PM, VD-0002) in Adult Subjects With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Collaborators: VioQuest Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14675; VQ-TCN-05-001 (Other: Vioquest)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2015-05

CONDITIONS: Cancer
Keywords: Phase I; Pharmacokinetics; TCN-PM; VD-0002; Immunohistochemistry; Serum tumor marker; Akt phosphorylation; Ex vivo testing; metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental): Phase I: Triciribine Phosphate Monohydrate
  Interventions: Drug: Triciribine Phosphate Monohydrate

INTERVENTIONS:
Drug: Triciribine Phosphate Monohydrate — 8 Cycles @ 28 days. Level 1: 15 mg/m^2; Level 2: 25 mg/m^2; 35 mg/m^2; 45 mg/m^2.
  Other Names: TCN-PM, BD-0002

SUMMARY:
Phase I dose escalation study of Triciribine Phosphate Monohydrate (TCN-PM) in patients with metastatic cancer whose tumors must be shown to be p-Akt positive. Study patients will be recruited from a Moffitt Cancer Center companion study (MCC-14474) "Immunohistochemical study of phosphorylated Akt in solid malignancies."

Each treatment cycle will consist of four weeks with TCN-PM being administered weekly (days 1, 8 and 15 every 28 days). Labs, vital signs (BP, HR, Resp Rate, Temp), and hematology and serum chemistry profile are to be performed weekly and/or prior to each treatment dose. Body Surface Area (BSA) should be calculated approximately every 8 weeks. Imaging studies (CT/MRI of chest, abdomen, and pelvis) and tumor response assessments will be performed every eight weeks or more frequently if indicated. Unless unacceptable toxicity occurs, the duration of treatment will be based on tumor reassessment.

DETAILED DESCRIPTION:
Phase I dose escalation study of Triciribine Phosphate Monohydrate (TCN-PM) in patients with metastatic cancer. Study patients will be recruited from a companion study [MCC-14474 "Immunohistochemical study of phosphorylated Akt in solid malignancies"], and potential subjects tumors' must be shown to be p-Akt positive.

Pretreatment evaluations are chest roentgenogram (CXR) and CT/MRI scans of the sites of known disease, performance status, tumor biopsy, MUGA (EF only), and a pregnancy test. A CT/MRI scan of the chest, abdomen, and pelvis known sites of disease is required at baseline and an immunohistochemical (IHC) assay for determination of akt expression (positive) prior to study drug administration.

Each treatment cycle will consist of four weeks with TCN-PM being administered weekly(days 1, 8 and 15 every 28 days). Labs, vital signs (BP, HR, Resp Rate, Temp), and hematology and serum chemistry profile are to be performed weekly and/or prior to each treatment dose. Body Surface Area (BSA) should be calculated approximately every 8 weeks. Imaging studies (CT/MRI of chest, abdomen, and pelvis) and tumor response assessments will be performed every eight weeks or more frequently if indicated.

Palliative and supportive care for other disease-related symptoms and for toxicity associated with treatment will be offered to all patients on this trial. Unless unacceptable toxicity occurs, the duration of treatment will be based on tumor reassessment done every eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Must consent to companion study MCC-14674 Immunohistochemical study of phosphorylated Akt in solid malignancies"
* Histologically documented cancer which is p-Akt positive by immunohistochemistry (IHC).
* Bi-dimensionally Measurable disease. If the only measurable disease is located in a previously irradiated area, definitive progression following irradiation must be documented.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 2 at study entry
* Adequate recovery from recent surgery, chemotherapy and radiation therapy. At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or prior radiation therapy.
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.
* Patients must be refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.
* Tumor site that is accessible to repetitive biopsies. Four core biopsies of the primary or metastatic tumor sites (or recurrence) are required prior to treatment initiation, and approximately 16 days after treatment initiation.
* Coagulation testing including Partial Thromboplastin Time (PTT), Prothrombin Time (PT), or International Normalization Ratio (INR) less than 1.5 times the upper limit of normal.
* Life expectancy of at least 3 months (12 weeks).
* Age greater than or equal to 18 years
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea greater than or equal to 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level greater than 35 mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG, or in accordance with local regulations, whichever is more sensitive) within 72 hours prior to the start of study medication or in accordance with local regulations, whichever is of shorter duration.

Exclusion Criteria:

* A baseline prolongation of QT/QTc interval >450 milliseconds (ms)
* A history of additional risk factors for torsades des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Dependent upon results of periodic testing
  To determine the dose of TCN-PM (VD-0002) (administered as a one-hour infusion days 1, 8, 15 every 28 days) which will inhibit by at least 50% Akt phosphorylation by ex vivo testing of tumor tissue samples

SECONDARY OUTCOMES:
Pharmacokinetics of TCN-PM,VD-0002 | Dependent upon results of periodic testing
  To characterize the pharmacokinetics of TCN-PM (VD-0002) when administered as a one-hour infusion days 1, 8 and 15 every 28 days
Radiologic response rate | Dependent upon results of periodic testing
  To monitor for drug efficacy, as determined by: radiologic response rate (RECIST criteria)
Biochemical response rate | Dependent upon results of periodic testing
  To monitor for drug efficacy, as determined by: biochemical response rate (if a serum tumor marker is present)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wenham, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Insitute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center website for clinical trials — http://www.moffitt.org